CLINICAL TRIAL: NCT06130085
Title: Open Labeled Randomized Clinical Trial of Introduction of a Partially Hydrolyzed Formula in Cow's Milk Protein Allergy After 6 Months of Elimination Protocol
Brief Title: Partially Hydrolyzed Formula in Cow's Milk Protein Allergy After 6 Months of Elimination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD444/2017
Record Dates: First submitted 2023-07-15; First posted 2023-11-13 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Cow's Milk Protein Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infants Continuing on amino acid based formula after 6 months elimination (No Intervention)
- Infants receiving partially hydrolyzed formula after 6 months of elimination diet (Active Comparator)
  Interventions: Dietary Supplement: Partially hydrolyzed formula

INTERVENTIONS:
Dietary Supplement: Partially hydrolyzed formula — Partially hydrolyzed formula given as the milk supplement for cow milk allergy patients after 6 months of strict elimination diet
  Arms: Infants receiving partially hydrolyzed formula after 6 months of elimination diet

SUMMARY:
For Patients diagnosed as cow milk protein allergy: Elimination of cow's milk products (CMPs) for 6 months.

All infants were supplemented with Amino Acid-based Formula (AAF) (Neocate infant®/ Neocate junior®, Dannone Nutricia) for 6 months at start of elimination diet.

For mixed milk fed infants (still receiving breast milk with the formula), mothers were encouraged to continue breast-feeding while avoiding all milk and milk products from their own diet.

Intervention after completing 6 months of eliminating CMPs. The included patients were randomly assigned to one of (2 groups).

1. Group I (AAF group) n= 50 Infants in this group continued with Amino Acid-based Formula for another 6 months.
2. Group II (pHF group) n= 50 Infants in this group were shifted gradually to Partially-hydrolyzed whey formula (pHF) (Liptomil Plus HA infant formula. for another 6 months with continuation of elimination of cow's milk products.

They were followed up for manifestations of intolerance to pHF. Infant who showed manifestations of intolerance were returned to AAF and continued for 6 months with AAF.

Final step: Reintoduction of CMPs After 12 months of elimination of CMPs, evaluation of tolerance to whole CMPs was done by oral food challenge (OFC).

For infants who were still non-tolerant to CMPs after 12 months of elimination were followed up and re-challenged after 6 months.

DETAILED DESCRIPTION:
Phase Ⅰ:Initial assessment at enrollment i. Full medical history taking: with emphasis on: Personal History: Age- Sex- Order of birth- Consanguinity-Residence

Main presenting symptoms:

A- Gastrointestinal symptoms: at initial diagnosis According to the clinical presentations, following clinical diagnoses were identified GERD, FPIAP, FPIES, FPE, constipation and combination of symptoms as shown in the following table.

B- Associated systemic allergic manifestations: at initial diagnosis C- CoMiSS: Cow's Milk-related Symptom Score (CoMiSS) at presentation. CMPA diagnosis was confirmed by an elimination diet followed by an oral food challenge.

D- Course of the disease:

E- Dietary and nutritional history:

1. Breast Feeding: If Yes exclusive for how long?
2. Artificial feeding: Age of start, type of formula, Indication.
3. Weaning: Time of start, Type of food given (each food and time of introduction especially cow's milk and CMPs), Any problems during weaning (gastrointestinal, respiratory or skin allergies) and eliciting dose of milk products that caused symptoms.
4. Accidental intake of raw or heated milk during elimination period and its consequences.

   * Past history: mode of delivery
   * Family history: atopy, siblings with CMPA
   * Medication history: Antireflux medications, laxatives, probiotics. ii. Clinical examination:
   * Anthropometric measurements: (weight &height on Z score, Wt/Ht ratio) using WHO 2006 Growth charts to those aged ≤ 2 years & CDC Growth charts 2000 if >2 years old
   * Signs of allergy: (atopic dermatitis- allergic rhinitis-wheezy chest)
   * Abdomen:(Distension- Tenderness- organomegaly)
   * Perineal area: (Perianal inflammation, napkin rash)

Phase 2: Elimination of CMPs for 6 months. All infants were supplemented with Amino Acid-based Formula (Neocate infant®/ Neocate junior®, Dannone Nutricia) for 6 months at start of elimination diet. Cow's-milk-based formula and supplementary foods containing CMPs, other animal milk proteins (eg, goat's milk, sheep's milk) were strictly avoided due to cross reactivity.

For mixed milk fed infants (still receiving breast milk with the formula), mothers were encouraged to continue breast-feeding while avoiding all milk and milk products from their own diet Breast feeding mothers excluding cow's milk were prescribed a supplement of 1000 mg of calcium & 10 µg (400 IU) of vitamin D every day

Phase III: Intervention after completing 6 months of eliminating CMPs

o The included patients were randomly assigned to one of (2 groups).

1. Group I (AAF group) n= 50 Infants in this group continued with Amino Acid-based Formula for another 6 months.
2. Group II (pHF group) n= 50 Infants in this group were shifted gradually the same way as OFC (from Amino Acid-based Formula; to Partially-hydrolyzed whey formula (Liptomil Plus HA infant formula; for another 6 months with continuation of elimination of CMPs.

They were followed up for manifestations of intolerance to pHF. Infant who showed manifestations of intolerance were returned to AAF and continued for 6 months with AAF.

Phase IV: Reintroduction of CMPs After 12 months of elimination of CMPs, evaluation of tolerance to whole CMPs was done by OFC. Tolerance was established by a negative challenge followed by regular ingestion of age-appropriate quantities of cow's milk at home without symptoms, where patients were followed up again for one month to detect any symptoms of intolerance after regular ingestion of milk products

For infants who were still non-tolerant to CMPs after 12 months of elimination were followed up and re-challenged after 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Artificially fed infants whether exclusively or complementary.
2. Confirmed diagnosis of CMPA based on clinical symptoms and signs and followed by withdrawal open re-challenge test

Exclusion Criteria:

1. Exclusively breast-fed infants.
2. Anaphylactic type.
3. Multiple food Allergies.

Ages: 7 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
compare the rate of tolerance to cow milk products among patients allocated to partially hydrolyzed formula after 6 months of milk free diet compared to those who completed 1 year of elimination | At the month 13 for both groups and for extra more 30 days of regular ingestion of cow's milk products
  Questionnaire done to assess occurrence of following symptoms Vomiting, Hematemesis, Diarrhea (using BRISTOL scale), Constipation, Eczema, Skin rash, Perianal inflammation, weight loss in kilograms or failure to gain weight in kilograms, (Colic, Straining and marked Abdominal distension), skin rash, angioedema, and recurrent respiratory symptoms within two months of following up after milk reintroduction. If any of the previous items is present, then the patient is considered intolerant to milk. All items should be answered by (no) in order to consider the patient tolerant to milk

SECONDARY OUTCOMES:
Tolerance to pHF after 6 months elimination diet | At the seventh month in the group allocated to receive pHF after six months of elimination diet
  To assess tolerance to partially hydrolsed milk formula in the group assigned to ingest pHF via a Questionnaire done to assess occurrence of following symptoms Vomiting, Hematemesis, Diarrhea (using BRISTOL scale), Constipation, Eczema, Skin rash, Perianal inflammation, weight loss in kilograms or failure to gain weight in kilograms, (Colic, Straining and marked Abdominal distension), skin rash, angioedema, and recurrent respiratory symptoms within two months of following up after milk reintroduction. If any of the previous items is present, then the patient is considered intolerant to milk. All items should be answered by (no) in order to consider the patient tolerant to pHF.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Vandenplas Y, Dupont C, Eigenmann P, Host A, Kuitunen M, Ribes-Koninckx C, Shah N, Shamir R, Staiano A, Szajewska H, Von Berg A. A workshop report on the development of the Cow's Milk-related Symptom Score awareness tool for young children. Acta Paediatr. 2015 Apr;104(4):334-9. doi: 10.1111/apa.12902. Epub 2015 Jan 29. PMID 25557474
- [Background] Nowak-Wegrzyn A, Chehade M, Groetch ME, Spergel JM, Wood RA, Allen K, Atkins D, Bahna S, Barad AV, Berin C, Brown Whitehorn T, Burks AW, Caubet JC, Cianferoni A, Conte M, Davis C, Fiocchi A, Grimshaw K, Gupta R, Hofmeister B, Hwang JB, Katz Y, Konstantinou GN, Leonard SA, Lightdale J, McGhee S, Mehr S, Sopo SM, Monti G, Muraro A, Noel SK, Nomura I, Noone S, Sampson HA, Schultz F, Sicherer SH, Thompson CC, Turner PJ, Venter C, Westcott-Chavez AA, Greenhawt M. International consensus guidelines for the diagnosis and management of food protein-induced enterocolitis syndrome: Executive summary-Workgroup Report of the Adverse Reactions to Foods Committee, American Academy of Allergy, Asthma & Immunology. J Allergy Clin Immunol. 2017 Apr;139(4):1111-1126.e4. doi: 10.1016/j.jaci.2016.12.966. Epub 2017 Feb 4. PMID 28167094
- [Background] Mehta NM, Corkins MR, Lyman B, Malone A, Goday PS, Carney LN, Monczka JL, Plogsted SW, Schwenk WF; American Society for Parenteral and Enteral Nutrition Board of Directors. Defining pediatric malnutrition: a paradigm shift toward etiology-related definitions. JPEN J Parenter Enteral Nutr. 2013 Jul;37(4):460-81. doi: 10.1177/0148607113479972. Epub 2013 Mar 25. PMID 23528324
- [Background] Luyt D, Ball H, Makwana N, Green MR, Bravin K, Nasser SM, Clark AT; Standards of Care Committee (SOCC) of the British Society for Allergy and Clinical Immunology (BSACI). BSACI guideline for the diagnosis and management of cow's milk allergy. Clin Exp Allergy. 2014;44(5):642-72. doi: 10.1111/cea.12302. PMID 24588904
- [Background] Ludman S, Shah N, Fox AT. Managing cows' milk allergy in children. BMJ. 2013 Sep 16;347:f5424. doi: 10.1136/bmj.f5424. No abstract available. PMID 24041704
- [Background] Lightdale JR, Gremse DA; Section on Gastroenterology, Hepatology, and Nutrition. Gastroesophageal reflux: management guidance for the pediatrician. Pediatrics. 2013 May;131(5):e1684-95. doi: 10.1542/peds.2013-0421. Epub 2013 Apr 29. PMID 23629618